CLINICAL TRIAL: NCT04142476
Title: Evaluation of the Impact of a Pharmaceutical Interview on the Adherence to Hormonotherapy in Women With Breast Cancer
Acronym: HORMONOVILLE
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: insufficient recruitment
Sponsor: Centre Georges Francois Leclerc (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: HORMONOVILLE
Record Dates: First submitted 2019-10-24; First posted 2019-10-29 (Actual); Last update posted 2025-02-17 (Actual); Status verified 2025-02

CONDITIONS: Breast Cancer
Keywords: Hormonotherpy; Compliance
MeSH Terms: conditions — Breast Neoplasms; Patient Compliance | interventions — Interviews as Topic

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Pharmaceutical Interview (Experimental): Pharmaceutical Interview to motivate patient in his hormonotherapy's compliance
  Interventions: Other: interview

INTERVENTIONS:
Other: interview — interviews with patient's pharmacist to motivate in the hormonotherapy's compliance.

SUMMARY:
Breast cancer is the first cancer in women and 60% of new cases occurring in women 50 to 74 years old. With about 50,000 new cases, it is the second cancer the most serious cancers. In the therapeutic strategy, hormone therapy takes pride of place by allowing a significant reduction in the recurrence rate.

For the hormonotherapy be effective, patient compliance should be optimal during treatment. Different factors or barriers may lead to a lack of adherence, such as the occurrence of adverse effects, treatment fatigue, a difficult relationship with the health care team, beliefs about success or the need for treatment.

In order to facilitate the compliance of hormonoherapy treatment by patients, it is important to include different health professionals such as pharmacists.

DETAILED DESCRIPTION:
Hormonotherapy adherence to breast cancer patients could be improved by :

* the use of electronic pill dispensers since the first prescription to visualize the level of compliance of each patient and study with her the various factors that can limit it.
* motivational, semi-directed and scheduled drug interviews at regular intervals throughout the study over a period of 18 months to visualize the compliance rate (ratio of the number of tablets taken by the patient on the number of tablets to be taken theoretically over the period), to evaluate the presence or absence of iatrogenesis specific to hormone therapy and to ensure adequate medical follow-up.

ELIGIBILITY:
Inclusion Criteria:

1. Woman, over 18 years old.
2. With non-metastatic breast cancer.
3. Treated by hormone therapy, regardless of the molecule (cancer RH positive).
4. In primary prescription of hormone therapy.
5. First prescription by a medical oncologist, surgeon or radiation therapist from the CGFL.
6. Pharmacy of the patient located in the perimeter defined in the context of the study (Residents in the Burgundy region between a triangle delimited by the towns of Chatillon sur Seine, Dole and Chalon sur Saone.
7. Woman who received information about the study and gave her written consent.
8. Affiliation to a social security scheme.
9. Participant Agreement of the referent city pharmacy of the patient.

Exclusion Criteria:

1. Metastatic patient.
2. Patient participating in another epidemiological or clinical study of adherence and / or hormone therapy.
3. Patient under guardianship, curatorship or safeguard of justice.
4. Patient with severe psychiatric disorders or who does not speak the French language
5. Refusal to participate in the study.
6. Refusal of participation of the referent city pharmacy of the patient.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 105 (Actual)
Dates: Start 2019-06-25 (Actual); Primary Completion 2023-02-07 (Actual); Study Completion 2023-02-07 (Actual)

PRIMARY OUTCOMES:
Patient compliance | 18 months
  data from electronic pillboxes

CONTACTS AND LOCATIONS:
Locations (1):
- Centre Georges Francois Leclerc, Dijon, France